CLINICAL TRIAL: NCT05399472
Title: Regional Interdependence Between Functional Hallux Limitus and Ankle Dorsiflexion in Healthy Adolescent Athletes
Brief Title: Teenage Functional Hallux Limitus and Ankle Dorsiflexion Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Ballardin Francesco, Clinical Professor, University of Bologna
Other Study IDs: TMUNIBO2022PS
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Hallux Limitus; Ankle Joint
Keywords: Functional hallux limitus; Ankle dorsiflexion
MeSH Terms: conditions — Hallux Limitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant: The participants must be teenage basketball players (12-17 years old).
  The exclusion criteria are:
  * have suffered in the last 3 months of lower limb musculoskeletal disorders such as pain for more than 7 days (ankle distortion outcomes, leg/foot fractures, plantar fasciopathy, metatarsalgias, etc);
  * athletes who have undergone surgery on their lower limb.
  Interventions: Diagnostic Test: Dorsiflexion lunge test; Diagnostic Test: Jack Test

INTERVENTIONS:
Diagnostic Test: Dorsiflexion lunge test — The dorsiflexion lunge test (DLT) will be used to measure ankle dorsiflexion. To perform this test, the participant stands in front of a wall holding the foot of their limb to be measured perpendicularly to it. The other foot is to be kept behind it. The participant is asked to perform a lunge (to dorsiflex the ankle and bring the knee into flexion) until the front knee touches the wall without the heel lifting off the ground. The participant steps away from the wall as much as possible as long as the knee keeps touching the wall. Measurement in centimeters is taken from the heel of the examined leg to the wall.
Diagnostic Test: Jack Test — The Jack Test will be used to measure the first toe dorsiflexion under load. The examiner pulled the proximal phalanx of the hallux to dorsiflexion with his hand until the maximal amount of mobility was reached with the subject standing. The static arm of the goniometer was placed along the first metatarsal longitudinal axis while the free movable arm followed the proximal phalanx of the hallux axes.

SUMMARY:
This study aims to identify a possible correlation between reduced mobility of the first toe under load and reduced mobility of the ankle ROM in healthy adolescent basketball players. To reach this goal, two non-invasive tests will be performed to measure the amount of movement of the ankle joint and the first toe.

DETAILED DESCRIPTION:
Functional hallux limitus (FHL) is a common condition of the first metatarsophalangeal joint (MTF) characterized by reduced dorsiflexion (DF) under load and has a negative effect on load transfer during toe off.

This condition is especially common among athletes, even at a youth age, due to repeated loads that can lead to tissue and/or joint damage. The compensations that occur in athletes with an FHL can negatively affect sports performance and start injuries.

Limited ankle dorsiflexion under load is another element that can affect sports performance as well as predisposing to injury. Several studies have investigated its regional interdependence but only a few have hypothesized a correlation between this limitation and FHL.

The aim of this study is to understand a possible correlation between reduced ankle DF and reduced MTF dorsiflexion during loading, so that preventive action can be taken to reduce the risk of injury.

Participants will fill in a cross-check survey to establish if there are any predisposing factors for FHL or ankle DF reduction.

The dorsiflexion lunge test (DLT) will be used to measure ankle dorsiflexion. The Jack Test will be used to measure first toe dorsiflexion under load and the Dorsiflexion Lunge Test will be used to measure ankle DF.

ELIGIBILITY:
Inclusion Criteria:

* male teenages basketball players enrolled in a competitive sports club
* teenagers whose parents have signed the privacy and consent forms

Exclusion Criteria:

* athletes who have suffered in the last 3 months of lower limb musculoskeletal disorders such as pain for more than 7 days (ankle distortion outcomes, leg/foot fractures, plantar fasciopathy, metatarsalgias, etc);
* athletes who have undergone surgery on their lower limb.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Male teenager basketball players from Bologna competitive sports clubs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Dorsiflexion Lunge Test | T1: first day
  Measurement in centimeters taken from the heel of the examined leg to the wall.
Jack test | T1: first day
  Degrees of movement will be measured with a goniometer. Static arm of the goniometer was placed along the first metatarsal longitudinal axis while the free movable arm followed the proximal phalanx of the hallux axes.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Study Director — Università degli studi di Bologna; Silvia Pozzan, Principal Investigator — Università degli studi di Bologna; Tommaso Torriglia, Study Chair — Università degli studi di Bologna
Locations (1):
- Dipartimento di scienze biomediche e Neuromotorie (DIBINEM) - Università di Bologna (MED/48), Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be sharing by a publication and will be stored and shared with those who request it while maintaining the anonymity of participants.

REFERENCES:
- [Background] Payne C, Chuter V, Miller K. Sensitivity and specificity of the functional hallux limitus test to predict foot function. J Am Podiatr Med Assoc. 2002 May;92(5):269-71. doi: 10.7547/87507315-92-5-269. PMID 12015407
- [Background] Van Gheluwe B, Dananberg HJ, Hagman F, Vanstaen K. Effects of hallux limitus on plantar foot pressure and foot kinematics during walking. J Am Podiatr Med Assoc. 2006 Sep-Oct;96(5):428-36. doi: 10.7547/0960428. PMID 16988174
- [Background] Lafuente G, Munuera PV, Dominguez G, Reina M, Lafuente B. Hallux limitus and its relationship with the internal rotational pattern of the lower limb. J Am Podiatr Med Assoc. 2011 Nov-Dec;101(6):467-74. doi: 10.7547/1010467. PMID 22106194
- [Background] Durrant B, Chockalingam N. Functional hallux limitus: a review. J Am Podiatr Med Assoc. 2009 May-Jun;99(3):236-43. doi: 10.7547/0980236. PMID 19448175
- [Background] Aranda Y, Munuera PV. Plantar fasciitis and its relationship with hallux limitus. J Am Podiatr Med Assoc. 2014 May;104(3):263-8. doi: 10.7547/0003-0538-104.3.263. PMID 24901585
- [Result] Sanchez-Gomez R, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Calvo-Lobo C, Navarro-Flores E, Palomo-Lopez P, Romero-Morales C, Lopez-Lopez D. Reliability Study of Diagnostic Tests for Functional Hallux Limitus. Foot Ankle Int. 2020 Apr;41(4):457-462. doi: 10.1177/1071100719901116. Epub 2020 Jan 29. PMID 31994419
- [Result] Tregouet P. An assessment of hallux limitus in university basketball players compared with noncompetitive individuals. J Am Podiatr Med Assoc. 2014 Sep-Oct;104(5):468-72. doi: 10.7547/0003-0538-104.5.468. PMID 25275734
- [Result] Hall C, Nester CJ. Sagittal plane compensations for artificially induced limitation of the first metatarsophalangeal joint: a preliminary study. J Am Podiatr Med Assoc. 2004 May-Jun;94(3):269-74. doi: 10.7547/0940269. PMID 15153589